CLINICAL TRIAL: NCT05807555
Title: Longitudinal Evolution of Biomarkers of Dysautonomia and Inflammation During Sepsis in Children - An Observational Study
Brief Title: Longitudinal Evolution of Biomarkers of Dysautonomia and Inflammation During Sepsis in Children
Acronym: DysREAped
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 22CH528; 2022-A02587-36 (Other: ANSM)
Record Dates: First submitted 2023-02-13; First posted 2023-04-11 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Sepsis; Autonomic Nervous System
Keywords: Dysautonomia
MeSH Terms: conditions — Sepsis; Autonomic Nervous System Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infant with sepsis (Case): Patient hospitalized in the pediatric intensive care unit (ICU) for severe sepsis
  Interventions: Other: Ambulatory ECG; Biological: Blood sample
- Healthy child of the same sex and age (Control): Healthy children will be matched to cases by age and gender
  Interventions: Other: Ambulatory ECG

INTERVENTIONS:
Other: Ambulatory ECG — 24h ECG monitoring
Biological: Blood sample — The usual biological tests necessary for the management of the child and the addition of 1 tube of 2 ml
  Groups: Infant with sepsis (Case)

SUMMARY:
The Autonomic Nervous System (ANS) regulates the inflammatory response in real time, just as it controls heart rate and other vital functions.

Many studies have investigated induced stimulation of the vagus nerve and its therapeutic effect in inhibiting TNFα (Tumor Necrosis Factor alpha) secretion, and therefore the risk of hypotension, septic shock, organ dysfunction during inflammation.

While the anti-inflammatory effect of the autonomic nervous system on inflammation has been well studied, conversely, the effect of major inflammation on the balance of the autonomic nervous system is more difficult to understand. The inflammatory reflex could be overwhelmed and the regulatory centers of the brainstem dysregulated during situations of extreme inflammation.

DETAILED DESCRIPTION:
The purpose of this study is to follow the short-term evolution of sympathetic and parasympathetic markers of dysautonomia in children hospitalized in intensive care units for severe sepsis, to characterize the evolution of the different autonomic indices according to the site of infection (meningitis, pulmonary infection, organ failure, bacteraemia) and types of pathogens (viral, bacterial, atypical germs) and correlating the evolution of the various inflammation biomarkers and cytokines with the degree of dysautonomia.

ELIGIBILITY:
Inclusion Criteria for cases group :

* Hospitalization in a pediatric intensive care unit.
* Presenting the sepsis criteria
* Patient affiliated or entitled to a social security scheme
* Holders of parental authority having received informed information about the study and having signed the consent form

Exclusion Criteria for cases group :

* Parents or legal guardians who do not speak French
* Chronic or acute pathology that can alter autonomic balance (congenital heart disease, encephalopathy, neuropathy, acute pain, etc.)
* Recent general anesthesia less than 48 hours old. (inclusion may be made beyond 48 hours from the last general anesthesia if the inclusion criteria remain present)
* Taking treatments that can alter the ANS (β-blockers, etc.) or inflammation (NSAIDs, corticosteroids)

Inclusion criteria for control group :

* Patient affiliated or entitled to a social security scheme
* Holders of parental authority having received informed information about the study and having signed the consent form

Exclusion Criteria for control group :

* Parents or legal guardians who do not speak French
* Chronic or acute pathology that can alter autonomic balance (congenital heart disease, encephalopathy, neuropathy, acute pain, etc.)
* Recent general anesthesia less than 1 month.
* Taking treatments that can alter the ANS (β-blockers, etc.) or inflammation (NSAIDs, corticosteroids)

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children hospitalized in pediatric intensive care unit for severe sepsis
  Healthy children
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Kinetic of the HF(High Frequency) index (ms2/Hz) of heart rate variability | Through discharge from the ICU, an average of 15 days
  Measure of the HF index of heart rate continuously at the patient's bed, during a quiet sleep phase at night, day by day for the entire duration of hospitalization in the ICU.

SECONDARY OUTCOMES:
Global activity indices (SDNN (Standard deviation of the NN (R-R) intervals) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Plot (Poincaré plot)) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Parasympathetic indices (pNN50 (Percentage of successive RR intervals that differ by more than 50 ms) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Parasympathetic indices RMSSD (Root mean square of successive RR interval differences) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Parasympathetic indices HF (High Frequency) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Sympathetic indices (LF, LF/HF ratio) evaluation | Through discharge from the ICU, an average of 15 days
  Measured continuously in quiet sleep at night, by temporal, geometric, frequency, fractal and entropy analysis
Evolution of biological markers of inflammation: CRP (C-reactive protein) (mg/L) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Procalcitonin (ng/mL) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Leukocytes (G/L) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Ferritin (µg/L)s | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Fibrinogen (g/L) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Platelets (G/L) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Evolution of biological markers of inflammation : Triglycerides (g/L) | Day : 1, at discharge from the ICU, an average of 90 days
  Collection of blood sampling for analysis
Interferon alpha, interferon beta and interferon gamma. | Day : 1, at discharge from the ICU, an average of 90 days
  Analysed by Luminex from blood sample (pg/mg)
Tumor Necrosis Factor (TNF) | Day : 1, at discharge from the ICU, an average of 90 days
  Analysed by Luminex from blood sample (pg/ml)
Interleukines (IL1, IL2, IL3; IL4, IL5, IL6, IL7, IL8, IL9, IL10, IL11, IL12, IL13) | Day : 1, at discharge from the ICU, an average of 90 days
  Analysed by Luminex from blood sample (pg/ml)
Presence or absence of virus in blood | Day : 1, at discharge from the ICU, an average of 90 days
  PCR (Polymerase chain reaction) multiplex
Presence or absence of bacteria in blood | Day : 1, at discharge from the ICU, an average of 90 days
  Blood cultures
Presence or absence of bacteria in bone-marrow | Day : 1, at discharge from the ICU, an average of 90 days
  Lumbar puncture
Presence or absence of bacteria in urine | Day : 1, at discharge from the ICU, an average of 90 days
  cytobacteriological examination of urine

CONTACTS AND LOCATIONS:
Overall Officials: HUGUES PATURAL, MD-PHD, Principal Investigator — CHU DE SAINT-ETIENNE
Locations (1):
- Chu de Saint-Etienne, Saint-Etienne, France